CLINICAL TRIAL: NCT06247111
Title: Post-Emergency Department Discharge Clinic Telehealth Program for Patients With Uncontrolled Hypertension: a Pilot Study
Brief Title: Monitoring Blood Pressure at Home
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lama Ghazi, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012428; P50MD017338 (NIH)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Placebo Comparator): Participants receive usual care from providers to manage their blood pressure
  Interventions: Other: Usual care
- Remote Blood Pressure Monitoring + Telehealth (Active Comparator): Participants will undergo remote blood pressure monitoring and pharmacist led telehealth intervention for blood pressure management
  Interventions: Other: Remote Blood Pressure Monitoring + Telehealth

INTERVENTIONS:
Other: Remote Blood Pressure Monitoring + Telehealth — Remote blood pressure monitoring and pharmacist led telehealth intervention for blood pressure management
  Arms: Remote Blood Pressure Monitoring + Telehealth
Other: Usual care — Participants receive usual care, no intervention.
  Arms: Usual Care

SUMMARY:
The overall goal of this project is to determine if measuring blood pressure at home and staying in contact with a team of pharmacists and physicians to manage your blood pressure is feasible. The study will enroll 24 participants at UAB who are seen at the Emergency Department Post-Discharge Clinic. Half of the participants (12 patients) will be asked to measure their blood pressure at home, and half of the participants (12 patients) will continue to receive usual care. Participants who measure their blood pressure at home will also meet with a pharmacist weekly over the phone to discuss blood pressure readings and have blood pressure medications prescribed if needed. This program will last 3 months.

DETAILED DESCRIPTION:
For all participants:

1. Participants will receive information on the importance of measuring blood pressure and ways to improve blood pressure.
2. Participants will complete questionnaires describing current socioeconomic position, medical history and healthcare needs.
3. Participants will come in for one research clinic visit to get blood pressure measured 3 months after enrollment in this study.

For participants asked to measure blood pressure at home:

1. Measure blood pressure twice a day at home, following the instructions provided. The study will provide participants with the device and send text message reminders each week day. Participants will return the device at study visit 3 months from now.
2. Following the instructions provided, participants will talk to a pharmacist over the phone weekly to discuss blood pressure and medications. All medication changes will be discussed with a collaborating physician.
3. Participants will complete questionnaires on satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at the Emergency Department Post-Discharge Clinic
* >=18 years
* Blood pressure >=130/80 mmHg and <=160/100 mmHg
* English speakers
* Have a smartphone

Exclusion Criteria:

* Patients with blood pressure >=160 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Total number of recruited participants | 2 years
  Measuring number of eligible participants that enroll in the study

CONTACTS AND LOCATIONS:
Overall Officials: Lama Ghazi, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No